CLINICAL TRIAL: NCT02986685
Title: The Clinical Efficacy and Safety of Trimebutine Maleate Combined With Rabeprazole in Patients With Grade A or B Reflux Esophagitis Whose Symptoms Refractory to Rabeprazole
Brief Title: Trimebutine Maleate Combined With Rabeprazole in Patients With Grade A or B Reflux Esophagitis Whose Symptoms Refractory to Rabeprazole
Acronym: rRE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funds
Sponsor: Xijing Hospital of Digestive Diseases (Other)
Collaborators: Ankang City Central Hospital (Other); Shaanxi Provincial People's Hospital (Other); Baoji Central Hospital (Other); Hanzhong Central Hospital (Other)
Responsible Party: Principal Investigator, Yongquan Shi, Professor of Digestive Diseases, Xijing Hospital of Digestive Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY-20162096-1
Record Dates: First submitted 2016-11-23; First posted 2016-12-08 (Estimated); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Refractory Reflux Esophagitis
Keywords: Refractory reflux esophagitis; Rabeprazole; trimebutine maleate
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Trimebutine; Rabeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trimebutine maleate + rabeprazole (Experimental): trimebutine maleate 200mg three times daily combined with rabeprazole 20mg once daily
  Interventions: Drug: Trimebutine Maleate; Drug: rabeprazole
- rabeprazole (Other): rabeprazole 20mg once daily
  Interventions: Drug: rabeprazole

INTERVENTIONS:
Drug: Trimebutine Maleate — Rabeprazole 20mg once daily was administered during the 8 weeks' screening stage ,then oral trimebutine maleate 200mg three times daily combined with rabeprazole 20mg once daily were administered to the experimental arm for 4 weeks.
  Arms: trimebutine maleate + rabeprazole
Drug: rabeprazole — Rabeprazole 20mg once daily was administered during the 8 weeks' screening stage,and rabeprazole 20mg once daily was administered to other arm for additional 4 weeks.

SUMMARY:
The research aims to investigate whether trimebutine maleate combined with rabeprazole can improve the clinical efficacy in patients With refractory Los Angeles grade A or B reflux esophagitis . A total of 500 patients with Grade A or B reflux esophagitis refractory to rabeprazole will be randomly divided into two groups.One will continue to receive rabeprazole treatment,and the other group will receive extra oral trimebutine maleate 200 mg three times daily for 4 weeks. The end of the study for every patient is the improvement of main symptoms. The primary and secondary analyses are the main symptoms score, endoscopy results, Gastroesophageal reflux disease questionnaire（GerdQ) score,Hospital Anxiety and Depression Scale(HADS) score, Athens insomnia scale and World Health Organization Quality of Life-Bref(WHOQOL-BREF)scale scores at the baseline and final assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with typical symptoms of heartburn sensation, or acid regurgitation,or both for at least 6 months.The symptoms were moderate or severe and at least three days a week in 7 days prior to the enrollment,which can complicate with Atypical and extraesophageal symptoms .
2. Diagnosed by upper gastrointestinal endoscopy within one month before enrollment with grade A or B reflux esophagitis according to Los Angeles classification

Exclusion Criteria:

1. History of endoscopic anti-reflux surgery,Fundoplication and major gastrointestinal surgery.
2. History of the chest or abdominal radiotherapy.
3. History of grade C or D reflux esophagitis,other gastrointestinal diseases such as Barrett's esophagus,zollinger-ellison syndrome, gastric or duodenal ulcer(excluding ulcer scar),large (>5cm)hiatus hernia,malignant tumor,esophageal stricture,esophageal and gastric Varices,hemorrhage or perforation of the digestive tract,mechanical ileus,et al.
4. The presence of serious comorbidities (liver, gallbladder, pancreas, spleen,kidney,heart,lung,blood system,endocrine,mental disease,autoimmunity and metabolic disorders) and malignant tumor of other organs.
5. Diagnosis of endocrine,neurological and autoimmunity disorders that may seriously affect motility(e.g. scleroderma or gastroparesis),and the primary esophageal motility disorders(achalasia,esophagospasm or nutcracker oesophagus).
6. Pregnancy or lactation during the study and follow-up period.
7. Use of antisecretory drugs(PPIs or H2RA),eradication of H pylori,drugs influenced the gastrointestinal motility,anticholinergics ,antipsychotics and so on within 4 weeks before the study.
8. Contraindications to trimebutine maleate or rabeprazole.
9. Use of drugs have interaction with the study drugs （e.g. cisapride ,procainamide, clopidogrel or ciclosporin),or drugs which may affect the results of the study(e.g. antisecretory drugs(PPIs or H2RA),prokinetics,mucosal protective drugs or anticholinergics),or drugs absorbed depending on the acidity of the gastric fluid(e.g.ketoconazole or digoxin),or CYP3A4,CYP2C19 inhibitors during the study.
10. Patients inability or refuse to consent, unable to complete the questionnaire,and have poor compliance to the treatment.
11. patients participated in other clinical trial 3 months before the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2017-10 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The change of main symptom （heartburn，acid regurgitation，non-cardiac chestpain，hoarseness，et，al）score from baseline to the end of 8 weeks | baseline ，the end of 8 weeks
  After the screening,the investigators defined the patients with main symptom score improvement less than 50% as the refractory reflux esophagitis patients.
  The results before and after treatment will be compared.
The change of main symptom （heartburn，acid regurgitation，non-cardiac chestpain，hoarseness，et，al）score from the end of 8 weeks to the end of 12 weeks | the end of 8 weeks ， the end of 12 weeks

SECONDARY OUTCOMES:
change of GerdQ score from baseline to the end of 8 weeks | baseline，the end of 8 weeks
  The results before and after treatment will be compared
change of GerdQ score from the end of 8 weeks to the end of 12 weeks | the end of 8 weeks，the end of 12 weeks
  The results before and after treatment will be compared
change of Athens insomnia scale score from baseline to the end of 8 weeks | baseline，the end of 8 weeks
  Athens insomnia scale score was used to evaluate the quality of sleep. The results before and after treatment will be compared
change of Athens insomnia scale score from the end of 8 weeks to the end of 12 weeks | the end of 8 weeks，the end of 12 weeks
  Athens insomnia scale score was used to evaluate the quality of sleep. The results before and after treatment will be compared
change of WHOQOL-BREF score from baseline to the end of 8 weeks | baseline ， the end of 8 weeks
  The quality of life for the refractory reflux esophagitis patients was assessed with the WHOQOL-BREF.The results before and after treatment will be compared
change of WHOQOL-BREF score from the end of 8 weeks to the end of 12 weeks | the end of 8 weeks， the end of 12 weeks
  The quality of life for the refractory reflux esophagitis patients was assessed with the WHOQOL-BREF.The results before and after treatment will be compared
change of HADS score from baseline to the end of 8 weeks | baseline，the end of 8 weeks
  Depression and anxiety was assessed with HADS.The results before and after treatment will be compared
change of HADS score from the end of 8 weeks to the end of 12 weeks | the end of 8 weeks , the end of 12 weeks
  Depression and anxiety was assessed with HADS.The results before and after treatment will be compared
change of the results of upper gastrointestinal endoscopy from baseline to the end of 12 weeks | baseline,the end of 12 weeks
  If the patients complete the upper gastrointestinal endoscopy before and after the treatment,the results of the mucosal healing will be analyzed.
The dietary habits of the patients with refractory Los Angeles class A or B reflux esophagitis | baseline
The comorbidities（e.g.,hypertension，chronic kidney disease，diabetes，IBS,Functional dyspepsia,et，al） of the patients with refractory Los Angeles class A or B reflux esophagitis | baseline
the smoking and alcohol drinking habits of the patients with refractory Los Angeles class A or B reflux esophagitis | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data for all primary and secondary outcome measures will be made available within 6 months of study completion